CLINICAL TRIAL: NCT06930040
Title: Effect of Action Observation Therapy Versus Kinesio Taping on Upper Extremity Function In Children With Erb's Palsy
Brief Title: Effect of Action Observation Therapy Versus Kinesio Taping on Upper Extremity Function In Children With Erb' Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Hassan mansour Abdelsalam Elhawary, Physiotherapist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-324
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Upper Extremity Function In Childern With Erb's Palsy
Keywords: Action Observation Therapy; Kinesio Taping; upper extremity function; Erb's Palsy

STUDY DESIGN:
Intervention Model Description: The examined group got 30 minutes of a standard, selected physical therapy program in addition to 30 minutes of AOT on the upper limb (total session time: 1 hour), 3 sessions per week for three consecutive months (total therapy time: 3 hours/week). g the excAction observation was executed with therapist guidance and repeated practice (3 repetitions for each task).
  Kenisiotaping :Shoulder taping will done using two Kinesiotex tapes(2.5 · 7 cm), in the form of I shape. The tapes follow the line of pull of the anterior and posterior deltoid muscle fibers applied in order to assist the deltoid muscle action .
  The tape was applied with the child in a sitting position by assistance from his care giver, while the therapist supported the child's arm.
Who Masked: Participant
Masking Description: The participants will not know the details of the intervention of the other groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment protocol in Group A ,Action observation therapy (Active Comparator): The examined group got 30 minutes of a standard, selected physical therapy program in addition to 30 minutes of AOT on the upper limb (total session time: 1 hour), 3 sessions per week for three consecutive months (total therapy time: 3 hours/week). Action observation was executed with therapist guidance and repeated practice (3 repetitions for each task). The child has been requested to perform the watched task with the same tool after observing a 3-minute video for each task on an adjustable monitor screen positioned one meter in front of him or her from forward, sideways, and backward directions. The therapist sat beside the child to provide verbal comments during the excursion and to guide the child's movement. The AOT for the examined group included six unimanual tasks and six bimanual tasks.
  Interventions: Other: Action observation therapy protocol
- Treatment protocol in Group B , Kenisiotaping (Active Comparator): Shoulder taping will done using two Kinesiotex tapes(2.5 · 7 cm), in the form of I shape. The tapes follow the line of pull of the anterior and posterior deltoid muscle fibers applied in order to assist the deltoid muscle action .
  The tape was applied with the child in a sitting position by assistance from his care giver, while the therapist supported the child's arm. The first tape was initiated from the upper border of the lateral 1/3 of the clavicle (origin of anterior fibers of the deltoid) to the deltoid prominence on the middle of the lateral side of the body of the humerus moving backward and lateralward while the arm was externally rotated and horizontally abducted.
  Interventions: Other: Kenisiotaping

INTERVENTIONS:
Other: Action observation therapy protocol — The examined group got 30 minutes of a standard, selected physical therapy program in addition to 30 minutes of AOT on the upper limb (total session time: 1 hour), 3 sessions per week for three consecutive months (total therapy time: 3 hours/week). Action observation was executed with therapist guidance and repeated practice (3 repetitions for each task). The child has been requested to perform the watched task with the same tool after observing a 3-minute video for each task on an adjustable monitor screen positioned one meter in front of him or her from forward, sideways, and backward directions. The therapist sat beside the child to provide verbal comments during the excursion and to guide the child's movement. The AOT for the examined group included six unimanual tasks and six bimanual tasks. The unimanual tasks included pressing a rubber stamp, stacking cups, drinking water from a cup, grabbing a pen, flipping cards, and putting things on a stick.
  Arms: Treatment protocol in Group A ,Action observation therapy
Other: Kenisiotaping — Shoulder taping will done using two Kinesiotex tapes(2.5 · 7 cm), in the form of I shape. The tapes follow the line of pull of the anterior and posterior deltoid muscle fibers applied in order to assist the deltoid muscle action .
  The tape was applied with the child in a sitting position by assistance from his care giver, while the therapist supported the child's arm. The first tape was initiated from the upper border of the lateral 1/3 of the clavicle to the deltoid prominence on the middle of the lateral side of the body of the humerus moving backward and lateralward while the arm was externally rotated and horizontally abducted. The second tape was initiated from the lower lip of the posterior border of the spine of the scapula towards also the humeral deltoid prominence moving forward and lateralward while the arm was horizontally adducted and internally rotated as if reaching to the outside of the contralateral hip.
  Arms: Treatment protocol in Group B , Kenisiotaping

SUMMARY:
The purpose of this study is to study the Effect of Action Observation Therapy versus Kinesiology Taping on upper extremity function In Erb's Palsy Children.

DETAILED DESCRIPTION:
Erb's palsy is a form of brachial plexus injury in which there is paralysis of the upper arm and shoulder girdle muscles due to an injury to the roots of 5th and 6th cervical roots or the upper part of the brachial plexus. It can also affect the feeling (sensation) in the arm.

Erb's palsy is otherwise known as Erb - Duchenne palsy. The incidence ranges globally from 0.2% to 0.4 %of live births. According to the World Health Organization, prevalence is generally 1-2% world- wide, with the higher numbers being in underdeveloped countries. Duchenne- Erb type constitutes a major form among brachial plexus palsied children as it accounts about 80-90% of all brachial plexus palsied cases as a result of unilateral upper trunk lesion. Erb's Palsy affects the nerves of the neck that control the motions of the arm. This condition turns muscles inward toward the body, disturbing mobility . It can occur during normal delivery if a baby's neck is stretched unnaturally as the head and shoulders pass through the birth canal. Early bodily trauma in the first few months of life may also lead to the palsy. Nearly all children recover completely, but occasionally there is some persistent nerve damage. It is important that some physiotherapy exercises are started early, which aim to prevent the arm becoming fixed in an abnormal position and improve the chances of a full recovery. The name of erb's palsy is derived from the doctor who first documented the condition. The word palsy refers to the weakness in the muscle- not paralysis. Erb's palsy symptoms have been improving or else it clears up on their own. While most of the cases are mild, each child will have various reactions to their nerve damage. Therefore, each child may require different kinds of intervention .

Erb's palsy is the affecting the muscles of the Early treatment may entail physical and occupational therapy, daily passive range of motion exercise, splinting to lessen the severity of biceps/triceps co-contraction. However, many times, deformations occur that require surgical intervention

The role of Physiotherapy in erb's palsy, prevent your baby's muscles from becoming short, prevent your baby's joints becoming stiff, give your baby the feeling of normal movement, so that when their recovery begins, they will not have forgotten how to use their arm (remember those kicks and punches in the womb), continue to stimulate the feeling in your baby's arm.

Kinesiology Tape A very useful physiotherapeutic modality nowadays, if applied properly is the kinesiology tape, which is valuable adjunct to therapeutic rehabilitations .Kinesio tape is thin and elastic tape that can be extended up to 120 -140% of its original Height, this elasticity result in less mechanism constraints. It allows a partial to full range of motion for the applied muscles and joints with different pulling forces to skin, it can be used both muscles relaxation and to facilitate muscle contraction depending on its application, it associated with improvement of the proprioception, strength, and range of motion of multiple joints.

The application of Kinesio tape depends on goals of treatment, include position of the affected area and amount of pre- stretch applied to the tape. Specific cut shapes of Kinesio tape are designed to allow for optimal responses. An -X‖ strip, -Y‖ strip and -I‖ strip all seek various results. Several studies reported the effectiveness of Kinesio tape which reducing spasticity of muscles, enhancing the dynamic activities, and also improving extremity functions and repositioning. This study was to assess the effect of Kinesio tape of improving functional activity for erb's palsy children.

Action observation Therapy When someone observes an action, the Superior Temporal Sulcus in the temporal lobe sends information to describe the visual input, the mirror neuron system encodes this information to interpret the motor input and sends it back to the Superior Temporal Sulcus, which matches the sensory input of the desired movement with the visual information of the observed action.

The patient is asked to observe a real-life or a videotaped physical performance of another subject during Action Observation Therapy, after which the patient is required to imitate these movements.

ELIGIBILITY:
Inclusion criteria :

1. Their ages will be ranged from Five Years to Seven years in both sexes.
2. The infants with Erb's palsy (C5-C6).
3. Muscle tone within normal and muscle power within functional range.

Exclusion criteria:

Any participant has one or more of the followings will be excluded:

1. Children less than Five Years months or more than Seven years..
2. Shoulder subluxation or dislocation.
3. Children with congenital disease and serious medical disorder.
4. Children undergoing surgical treatment.
5. Complete sensory loss.
6. Shoulder subluxation or dislocation.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the grip strength | After 12 week
  Assessment of the grip strength by using Hand and Held Dynamometer
Jebsen Hand Function Test | After 12 week
  Measure hand function for activities of daily living. It has 7 items include: writing, turning over 3-by-5 inch cards, picking up small common objects, simulated feeding, stacking checkers, picking up large light objects and picking up large heavy object

CONTACTS AND LOCATIONS:
Locations (1):
- Hassan Elhawary, Kafr ash Shaykh, Cario, Egypt

IPD SHARING:
Plan to Share IPD: Undecided